CLINICAL TRIAL: NCT05879744
Title: A Phase 1, Open-label, Dose Escalation and Dose Expansion Study of CLN-978 in Patients With Relapsed/Refractory (R/R) B-cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: A Study of CLN-978 in Patients With Relapsed or Refractory (R/R) B Cell Non-Hodgkin Lymphoma (B-NHL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cullinan Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLN-978-001
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: NHL; NHL, Relapsed, Adult
Keywords: Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A Dose Escalation (Experimental): Patients with R/R B-NHL treated with CLN-978 in dose escalation cohorts
  Interventions: Drug: CLN-978
- Part B Dose Expansion (Experimental): Patients with R/R DLBCL, R/R FL and other R/R B-NHL treated with CLN-978 at a dose selected from the Part A Dose Escalation arm.
  Interventions: Drug: CLN-978

INTERVENTIONS:
Drug: CLN-978 — CD19xCD3 T cell engager

SUMMARY:
CLN-978-001 is a Phase 1, open-label, dose escalation and dose expansion study of CLN-978 in patients with Relapse/Refractory (R/R) B-cell Non-Hodgkin Lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) PS ≤ 2
* Documented diagnosis of one of the below CD19+ B-cell neoplasms according to WHO classification (Swerdlow et al., 2016) or WHO classification 2008:

  1. Diffuse large B-cell lymphoma - de novo or transformed
  2. High-grade B-cell lymphoma
  3. Primary mediastinal large B-cell lymphoma
  4. Follicular lymphoma
  5. Mantle cell lymphoma
  6. Marginal zone lymphoma (nodal, extranodal, or mucosa-associated)
* Relapsed, progressive, and/or refractory disease after at least 2 lines of therapy.
* For Part B expansion cohorts:

  1. Cohort B1: R/R DLBCL that has relapsed after at least 2 prior therapies including a CD20 monoclonal antibody and anthracycline.
  2. Cohort B2: R/R FL (grade 1-3a) that has relapsed after at least 2 prior therapies including CD20 monoclonal antibody and an alkylating agent.
  3. Cohort B3: Other R/R B-NHL.
* Measurable disease defined as ≥1 measurable nodal lesion (long axis >1.5 cm and short axis >1.0 cm) or ≥1 measurable extra-nodal lesion (long axis >1.0 cm) on computed tomography (CT) scan or magnetic resonance imaging (MRI) AND baseline fluorodeoxyglucose-positron emission tomography (FDG-PET) scan demonstrating positive lesion(s) compatible with CT- or MRI-defined anatomical tumor sites.
* Laboratory parameters including the following:

  1. Lymphocyte count < 5 x 10^9/L
  2. Platelet count ≥ 75 x 10^9/L
  3. Absolute neutrophil count ≥ 1.0 x 10^9/L; growth factor support allowed in cases of documented bone marrow involvement
  4. Hemoglobin ≥ 9 g/dL, with or without transfusion
  5. Creatinine clearance ≥ 45 mL/min
  6. Total bilirubin ≤ 1.5 × upper limit of normal (ULN), except patients with confirmed Gilbert's Syndrome
  7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN (unless attributed to hepatic involvement by lymphoma)

Exclusion Criteria:

* Primary CNS lymphoma or known CNS involvement by lymphoma at study screening
* Known past or current malignancy other than the inclusion diagnosis
* Known clinically significant cardiac disease
* Significant central nervous system disease
* Prior organ allograft
* Confirmed history or current autoimmune disorder or other disease requiring ongoing immune suppression
* Active Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), or known Human Immunodeficiency Virus (HIV) infection
* Live virus vaccines within 28 days of the first dose of CLN-978, during treatment, and until the end of last dose of CLN-978
* Known active, clinically significant bacterial, viral, fungal, mycobacterial, parasitic, or other infection, including coronavirus disease of 2019 (COVID-19) infection, at the time of enrollment or within 7 days of the first dose of CLN-978.
* Prior treatment with any of the following:

  1. Allogeneic HSCT
  2. Autologous HSCT within 30 days prior to the first dose of CLN-978
  3. Chimeric antigen receptor T cell therapy (CAR-T) within 30 days prior to the first dose of CLN-978
  4. Any investigational CD19 x CD3 T cell engager (TCE)
  5. Unconjugated CD19 monoclonal antibody ≤ 4 weeks prior to the first dose CLN-978
  6. Radio-conjugated or CD19 antibody-drug conjugate ≤ 12 weeks prior to the first dose CLN-978
  7. Investigational or standard of care monoclonal antibodies, chemotherapy, or other investigational agent ≤ 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of CLN-978
  8. Radiation therapy (XRT), with the exception of focal treatment for symptom control, ≤ 4 weeks of the first dose of CLN-978
* Woman of child-bearing potential who is pregnant, breast-feeding, or plans to become pregnant
* Male patients who plan to father a child or donate sperm within 120 days of last study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CLN-978 based on AEs, AESIs, and SAEs | 24 months
  Incidence and severity of adverse events (AEs)/adverse events of special interest (AESIs)/serious adverse events (SAEs); incidence of dose interruptions and delays
Define dose regimen for CLN-978 | 24 months
  Dose-limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Assess preliminary efficacy of CLN-978 by overall response in patients with selective histologies of R/R B-NHL | 24 months
  Overall response rate (ORR)
Assess preliminary efficacy of CLN-978 by complete response in patients with selective histologies of R/R B-NHL | 24 months
  Complete response (CR)
Assess preliminary efficacy of CLN-978 by duration of response in patients with selective histologies of R/R B-NHL | 24 months
  Duration of response (DOR)
Select PK parameters of CLN-978: AUC | 24 months
  Area under-the-concentration-time curve of CLN-978
Select PK parameters of CLN-978: Cmax | 24 months
  Maximum concentration of CLN-978
Select PK parameters of CLN-978: Half-life | 24 months
  Half-life of CLN-978
Immunogenicity of CLN-978 and potential impact on drug exposure | 24 months
  Incidence of anti-drug antibodies to CLN-978

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Texas Southwestern Medical Center, Dallas, Texas